CLINICAL TRIAL: NCT03714984
Title: The Efficacy of Pre-operative Educational Pelvic Floor Intervention on Urinary Continence in Patients Underwent Robotic Prostatectomy. A Randomized Clinical Trial
Brief Title: The Efficacy of Pre-operative Educational Pelvic Floor Intervention on Urinary Continence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IEO 818
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-06

CONDITIONS: Prostatectomy; Pelvic Floor Disorders
Keywords: Prostatectomy; Pelvic Floor Disorders; Robotic Surgical Procedures; rehabilitation
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Preoperative Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: Superiority trial with 1:1 allocation ratio, randomized with two-arm parallel group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre operative exercise (Experimental): The educational pelvic floor intervention group will receive one months before surgery a physiotherapy visit were will be explain to patients and care giver the pelvic floor anatomy and biomechanics and how perform the exercises to be follow at home focusing on pelvic muscles awareness and contraction. Patients and care giver will receive a daily exercise diary to fill at home and will be advised to follow the exercise program.
  Interventions: Other: Pre operative exercise
- Control group (Active Comparator): The control group will be just informed about the study protocol and will not receive any pre-operative intervention.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Pre operative exercise — After randomization participants will be allocated in two groups. The educational pelvic floor intervention group will receive two months before surgery a physiotherapy visit were will be explain to patients and care giver the pelvic floor anatomy and biomechanics and how perform the exercises to be follow at home focusing on pelvic muscles awareness and contraction.
  Arms: Pre operative exercise
Other: Control Group — The control group will be just informed about the study protocol and will not receive any pre-operative intervention.
  Arms: Control group

SUMMARY:
Prostate cancer is the most common type of cancer between male population and urinary incontinence (UI) is the most common of long-term sequelae. Nowadays, robotic prostatectomy became the surgery standard but there is still discrepant results regards the incidence of UI and there is a lack of studies about the use of pelvic floor rehabilitation in this population. Our study aims to assesses the efficacy of preoperative educational method in urinary incontinence after robotic prostatectomy.

DETAILED DESCRIPTION:
Prostate cancer is the most common type of cancer between male population, with 161,300 new cases a year in the USA and an incidence of 10% in Italy. Since many years surgery is the treatment of choice, both at an early stage and in advanced cases, but involves side effects. From the post-operative problem presents in literature, urinary incontinence (UI) is the most common of long-term sequelae and significantly affects the quality of life and the psychological aspect in the post-surgical period. The incidence of UI after prostatectomy surgery varies between 0.8% and 87% in the first 3 and 6 months and between 5% and 44.5% after 1 year. This variability depends on the UI definition and the type of measurement used, which are not homogeneous among the various studies in the literature. Evaluations that are not objective make it difficult to compare the results obtained, thus creating discrepancies.

To date, robotic prostatectomy is becoming the gold standard for its recognized greater accuracy when compared with the open surgery and laparoscopic procedure, with a reduced learning curve for operators and giving better post-surgical results. Progress technological aspects, such as the three-dimensional vision of the operative field, the macroscopic magnification and better image resolution, have made the robotic procedure a less invasive surgery with better functional outcomes. Despite these factors, UI is still present and in the majority of cases management is not completely evidence based. Moreover there is not yet a definite consensus regarding the predictive factors (age, disease stage, body weight, prostate volume and other comorbidities) in the incidence of the UI.

When patients presents UI diagnoses, the conservative intervention through the pelvic floor rehabilitation is recommended in an attempt to reduce the impact of this complication. Muscle strengthening and pelvic floor awareness after surgery are used for years in clinical practice with results widely documented in the literature, but their effectiveness in the pre-operative period, especially if after robotic surgery, has not yet been sufficiently studied. Currently, there are discrepant results mainly due to the type of rehabilitative methodology applied and the time of beginning the preoperative treatment. Our study tries to evaluate, through an objective and reproducible measurement, the efficacy of a preoperative educational method in urinary incontinence after robotic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age >= 40 <= 70 years old
* Body mass Index <= 27
* Indication of robotic prostate surgery
* Tumor with clinical stage T1 and T2.
* Extracapsular Extension Score <= 3, measured with magnetic resonance before surgery.

Exclusion Criteria:

* Pathologic T3 tumor with radiotherapy indication
* Previous prostate surgery
* Previous urinary incontinence.
* Metabolic disorder
* Central or peripheral neurologic disorders
* Inability to understand informed consent or to carry out the rehabilitation protocol autonomously.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Change in self-reported urinary continence | 1,3,6 months and 1 year after surgery
  Continence (completely dry patient) will be defined as the sum of no urinary leakage reported by the patient in his bladder diary

SECONDARY OUTCOMES:
The degree of urinary incontinence. | 1,3,6 months and 1 year after surgery
  Assesment of the degree of urinary incontinence based on a 24 hours pad test.
Quality of life instrument | 1,3,6 months and 1 year after surgery
  Assesment of quality of life using the The Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire.
Assesment of the post traumatic distress using the Impact of event Scale (IES). | 1,3,6 months and 1 year after surgery
  Scale range from 0 to 4 with lower values representing better outcomes
Assesment of the individual resilience with the resilience scale for adults (RSA). | 1,3,6 months and 1 year after surgery
  Scale range from 1 to 5 with lower values representing better outcomes
Assesment of the urinary status with the International Consultation on Incontinence (ICIQ) Questionnaire. | 1,3,6 months and 1 year after surgery
  Summed of sub scales range from 0 to 3, 0 to 6 and 1 to 10. Minimum score of 1 and maximum score of 19, with lower values representing better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Felipe Nevola Teixeira, PT, Principal Investigator — European Institute of Oncology
Locations (1):
- Istituto Europeo di Oncologia, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fossati N, Di Trapani E, Gandaglia G, Dell'Oglio P, Umari P, Buffi NM, Guazzoni G, Mottrie A, Gaboardi F, Montorsi F, Briganti A, Suardi N. Assessing the Impact of Surgeon Experience on Urinary Continence Recovery After Robot-Assisted Radical Prostatectomy: Results of Four High-Volume Surgeons. J Endourol. 2017 Sep;31(9):872-877. doi: 10.1089/end.2017.0085. Epub 2017 Jul 21. PMID 28732186
- [Background] Centemero A, Rigatti L, Giraudo D, Lazzeri M, Lughezzani G, Zugna D, Montorsi F, Rigatti P, Guazzoni G. Preoperative pelvic floor muscle exercise for early continence after radical prostatectomy: a randomised controlled study. Eur Urol. 2010 Jun;57(6):1039-43. doi: 10.1016/j.eururo.2010.02.028. Epub 2010 Mar 1. PMID 20227168
- [Background] Moore KN, Valiquette L, Chetner MP, Byrniak S, Herbison GP. Return to continence after radical retropubic prostatectomy: a randomized trial of verbal and written instructions versus therapist-directed pelvic floor muscle therapy. Urology. 2008 Dec;72(6):1280-6. doi: 10.1016/j.urology.2007.12.034. Epub 2008 Apr 2. PMID 18384853
- [Background] Burgio KL, Goode PS, Urban DA, Umlauf MG, Locher JL, Bueschen A, Redden DT. Preoperative biofeedback assisted behavioral training to decrease post-prostatectomy incontinence: a randomized, controlled trial. J Urol. 2006 Jan;175(1):196-201; discussion 201. doi: 10.1016/S0022-5347(05)00047-9. PMID 16406909